CLINICAL TRIAL: NCT05401955
Title: Effects of a Physical Therapy and Therapeutic Exercise Program in Graft-versus-host Disease (GVHD)
Brief Title: Physiotherapy and Therapeutic Exercise Program in Graft-versus-host Disease (GvHD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Vicente Rodríguez Pérez, Associate Professor, University of Salamanca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Interventional
Record Dates: First submitted 2022-05-12; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: GVHD,Acute; GVHD, Chronic
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Graft versus host disease Group (Experimental)
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — An adapted physical exercise protocol

SUMMARY:
Range of motion, antropometric measurements, quality of life questionnaire and 2 minutes walk test will be implemented as an initial assessment.

Physical exercise program will take 2 sessions a week for six months, and several follow-ups: before, during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Allogenic Transplantation patients with Graft versus host disease

Exclusion Criteria:

* Cognitive impairment
* Physical limitation from other pathologies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
SF36 Questionnaire | baseline and post-intervention (24 weeks)
  Quality of life
2 minutes walk test | baseline and post-intervention (24 weeks)
  walking for 2 minutes without rest
Hands strength | baseline and post-intervention (24 weeks)
  Dynamometer
Active range of motion | baseline and post-intervention (24 weeks)
  P-ROM. Active ROM will be compared with standard pictures (1-4 points for lower limb and 1-7 points for upper limb)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salamanca, Salamanca, Spain